CLINICAL TRIAL: NCT05356819
Title: The Value of Integrated Pulmonary Index Monitoring
Brief Title: The Value of Integrated Pulmonary Index Monitoring in Detecting Respiratory Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Hale Kefeli Celik, Principal Investigator, Anesthesiologist, Samsun Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GOKA/2020/16/6
Record Dates: First submitted 2022-04-13; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Monitored Anesthesia Care
Keywords: Integrated Pulmonary Index (IPI) monitoring; capnograph; endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopy (Other): Integrated Pulmonary Index (IPI) monitor will be applied to the patients, to provide numerical data obtained from the measurements of end-tidal carbon dioxide, respiratory rate, oxygen saturation measured by pulse oximetry (SpO2), and pulse rate.
  Patients were administered 2 mg midazolam as premedication for 5 minutes before the procedure and propofol 1-1.3 mg/kg bolus for sedation, followed by repeated doses (10-30 mg) according to the Ramsey sedation score. All patients were given 2 lt/min oxygen via nasal cannula during the procedure.
  Interventions: Device: Smart Capnography™, Microstream®

INTERVENTIONS:
Device: Smart Capnography™, Microstream® — patients monitored by capnograph

SUMMARY:
Integrated Pulmonary Index (IPI) is a tool that provides numerical values on a scale of 1-10 based on physiological parameters such as peripheral oxygen saturation (SpO2), pulse rate, respiratory rate, end-tidal carbon dioxide (ETCO2). It is a valuable monitor for sedation procedures and can provide early warning during cardiorespiratory derangements.The aim of the study is to determine whether the Integrated Pulmonary Index (IPI) detects changes in ventilation status early in patients undergoing gastrointestinal endoscopy under sedation, and to determine the risk factors affecting hypoxia and severe hypoxia.

DETAILED DESCRIPTION:
A single-center and retrospective study was conducted in 154 patients who underwent upper and lower gastrointestinal system endoscopy in the endoscopy unit between October 2018 and December 2019. Patients who were monitored by capnograph in addition to routine monitoring (ECG, noninvasive blood pressure and pulse oximetry monitoring) during the procedure in the endoscopy unit were included in the study.

Patients were administered 2 mg midazolam as premedication for 5 minutes before the procedure and propofol 1-1.3 mg/kg bolus for sedation, followed by repeated doses (10-30 mg) according to the Ramsey sedation score. All patients were given 2 lt/min oxygen via nasal cannula during the procedure. In pulse oximetry, oxygen saturation longer than 15 seconds was defined as less than 92% hypoxia, and below 85% was defined as severe hypoxia.

IPI value was measured with Smart Capnography™, Microstream® Integrated Pulmonary Index device. According to the capnographic information obtained from the patients and preserved in the capnograph disc memory, the planned findings in the study are as follows:

1. Number of hypoxic events observed in patients (SaO2 value below 92% over 15 seconds)
2. Number of severe hypoxic events observed in patients (SaO2 value below 85%)
3. Apnea episodes observed in patients (observation of a straight line longer than 15 seconds on the capnograph, absence of respiratory activity)
4. Time from apnea to development of hypoxia and severe hypoxia in patients who develop hypoxia and severe hypoxia following apnea
5. Time between IPI=1, IPI<7, EtCO2=0 and hypoxia and severe hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Patients monitored by capnograph
* ASA I-III
* Patients who underwent an elective endoscopic procedure

Exclusion Criteria:

* Patients who do not have capnograph monitoring or whose capnography records are missing
* Emergency endoscopic intervention (GIS bleeding, trauma, etc.)
* ASA IV-V
* Patients with pre-procedure SaO2 value below 90%, systolic blood pressure below 90 mmHg, heart rate below 50 beats/minute

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Integrated pulmoner index and puls oxymetry | From the time between first sedative medication administration to the end of the procedure.
  The number of hypoxic events observed in patients (SaO2 value below 92% over 15 seconds) and number of severe hypoxic events observed in patients (SaO2 value below 85%)

CONTACTS AND LOCATIONS:
Overall Officials: HALE KEFELİ ÇELİK, MD, Study Director — Samsun Research and Education Hospital
Locations (1):
- Samsun Research and Education Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Our data and statistical analysis of each investigated all parameter and data are available after the publication of the clinical study

REFERENCES:
- [Result] Dumonceau JM, Riphaus A, Aparicio JR, Beilenhoff U, Knape JT, Ortmann M, Paspatis G, Ponsioen CY, Racz I, Schreiber F, Vilmann P, Wehrmann T, Wientjes C, Walder B; NAAP Task Force Members. European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates, and the European Society of Anaesthesiology Guideline: Non-anesthesiologist administration of propofol for GI endoscopy. Endoscopy. 2010 Nov;42(11):960-74. doi: 10.1055/s-0030-1255728. Epub 2010 Nov 11. PMID 21072716
- [Result] Wehrmann T, Riphaus A. Sedation with propofol for interventional endoscopic procedures: a risk factor analysis. Scand J Gastroenterol. 2008 Mar;43(3):368-74. doi: 10.1080/00365520701679181. PMID 18938664
- [Result] Riphaus A, Wehrmann T, Kronshage T, Geist C, Pox CP, Heringlake S, Schmiegel W, Beitz A, Meining A, Muller M, von Delius S. Clinical value of the Integrated Pulmonary Index(R) during sedation for interventional upper GI-endoscopy: A randomized, prospective tri-center study. Dig Liver Dis. 2017 Jan;49(1):45-49. doi: 10.1016/j.dld.2016.08.124. Epub 2016 Sep 1. PMID 27671621
- [Result] Michael FA, Peveling-Oberhag J, Herrmann E, Zeuzem S, Bojunga J, Friedrich-Rust M. Evaluation of the Integrated Pulmonary Index(R) during non-anesthesiologist sedation for percutaneous endoscopic gastrostomy. J Clin Monit Comput. 2021 Oct;35(5):1085-1092. doi: 10.1007/s10877-020-00563-2. Epub 2020 Jul 30. PMID 32734356